CLINICAL TRIAL: NCT01453361
Title: Phase II Trial of FANG™ Autologous Tumor Cell Vaccine in Advanced Melanoma
Brief Title: Phase II FANG™ in Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision to pursue other indications
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL 114
Record Dates: First submitted 2011-08-10; First posted 2011-10-17 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Advanced Melanoma
Keywords: FANG; Melanoma; Vigil
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vigil™ Vaccine (Experimental): Autologous Vigil™ vaccine will be supplied by Gradalis, Inc. Patients will receive 1 x 10e7 cells via intradermal injection one day each month for a minimum maximum of 12 doses as long as subject is clinically stable.
  Interventions: Biological: Vigil™ Vaccine

INTERVENTIONS:
Biological: Vigil™ Vaccine
  Other Names: formerly known as FANG™

SUMMARY:
Preliminary studies with a variety of vaccines suggest target accessibility (potential immunogenicity) in a variety of solid tumors to immune directed approaches. In an effort to overcome limitations of immunostimulatory cancer vaccines, the investigators have designed a novel autologous vaccine to address inability to fully identify cancer associated antigens, antigen recognition by the immune system (i.e. antigen to immunogen), effector potency, and cancer-induced resistance. In an effort to overcome limitations of immunostimulatory cancer vaccines, the investigators designed a novel dual-modulatory autologous whole cell vaccine, Vigil™ (bi-shRNA furin and GMCSF Autologous Tumor Cell Vaccine), incorporating the rhGMCSF (recombinant human GMCSF) transgene and the bifunctional shRNAfurin (to block proprotein conversion to active TGFb1 and b2) to 1) address the inability to fully identify cancer associated antigens, 2) effect antigen recognition by the immune system (i.e. antigen to immunogen), 3) enhance effector potency, and 4) subvert endogenous cancer-induced immune resistance. The investigators have also completed the Phase I assessment of Vigil™ vaccine in 27 advanced solid tumor patients (1.0 x 10e7 or 2.5 x 10e7 cells/injection/month for a maximum of 12 vaccinations) who have not experienced any significant adverse effects following 131 vaccinations, including 4 patients with melanoma. Plasmid functionality, immune biomarker response, and preliminary evidence of anticancer activity have been observed. This is a Phase II study of intradermal autologous Vigil™ cancer vaccine (1.0 x 10e7 cells/injection; maximum of 12 vaccinations) in patients with stages IIIc and IV melanoma with biopsy accessible lesions to document blood and intratumoral immune responses and assess correlation with survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Stages IIIc and IV melanoma.
2. Has been informed of all alternative ≥ second-line therapies that are the current standard of care. If no conventional frontline therapy indicated or acceptable by patient, patient may participate after review by sponsor.
3. Clinically (medically) indicated procedure (i.e. biopsy of lesions of recurrent disease, palliative management via resection, thoracentesis, etc.) to collect viable tumor in sufficient quantity ("golf ball size" estimated weight ~ 30 grams, pleural and/or ascites fluid estimated volume ≥ 500mL) for vaccine processing.
4. Recovered to ≤ Grade 1 (excluding alopecia) from all clinically relevant toxicities related to prior therapies.
5. Patients will be allowed to participate following single prior CNS treatment with stereotactic radiotherapy whole brain irradiation and stable without steroid requirement for ≥2 months or following ≥2 prior CNS treatments with stereotactic radiotherapy whole brain irradiation and stable without steroid requirement for ≥4 months.
6. Patients must be off all "statin" drugs for ≥ 2 weeks prior to initiation of therapy.
7. Age ≥18 years.
8. ECOG performance status (PS) 0-1.
9. Estimated >4 month survival probability.
10. Normal organ and marrow function as defined below:

    Absolute granulocyte count ≥1,500/mm3 Absolute lymphocyte count ≥500/mm3 Platelets ≥100,000/mm3 Total bilirubin ≤2 mg/dL AST(SGOT)/ALT(SGPT) ≤2x institutional upper limit of normal Creatinine <1.5 mg/dL
11. Ability to understand and the willingness to sign a written informed consent document.
12. Negative pregnancy test.

Exclusion Criteria:

1. Surgery involving general anesthesia, chemotherapy, radiotherapy, steroid therapy, or immunotherapy within 4 weeks prior to entering the study. Collection of lumenal tissue must be avoided.
2. Patient must not have received any other investigational agents within 30 days prior to study entry.
3. Patients with known active or symptomatic brain metastases.
4. Patients with compromised pulmonary disease.
5. Short term (<30 days) concurrent systemic steroids ≤ 0.25 mg/kg prednisone per day (maximum 7.5 mg/day) and bronchodilators (inhaled steroids) are permitted; other steroid regimens and/or immunosuppressives are excluded. Patients requiring steroids following previous CNS radiation for metastatic disease are excluded.
6. Prior splenectomy.
7. Prior malignancy (excluding nonmelanoma carcinomas of the skin) unless in remission for 2 years.
8. Kaposi's Sarcoma.
9. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Patients who are pregnant or nursing.
11. Patients with known HIV.
12. Patients with chronic Hepatitis B and C infection.
13. Patients with uncontrolled autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2016-03-22 (Actual); Study Completion 2016-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Mary Crowley Cancer Research Center
Locations (1):
- Mary Crowley Cancer Research Centers, Dallas, Texas, United States

REFERENCES:
- [Background] Olivares J, Kumar P, Yu Y, Maples PB, Senzer N, Bedell C, Barve M, Tong A, Pappen BO, Kuhn J, Magee M, Wallraven G, Nemunaitis J. Phase I trial of TGF-beta 2 antisense GM-CSF gene-modified autologous tumor cell (TAG) vaccine. Clin Cancer Res. 2011 Jan 1;17(1):183-92. doi: 10.1158/1078-0432.CCR-10-2195. PMID 21208907
- [Background] Maples PB, Kumar P, Yu Y, Wang Z, Jay CM, Pappen BO, Rao DD, Kuhn J, Nemunaitis J, Senzer N: FANG Vaccine: Autologous Tumor Cell Vaccine Genetically Modified to Express GM-CSF and Block Production of Furin. BioProcessing Journal 2010; 8(4):4-14.
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- See also: Follow-up of bi-shRNAfurin /GM-CSF Engineered Autologous Tumor Cell (EATC) Immunotherapy Vigil in patients with advanced melanoma — http://www.oatext.com/pdf/BGG-1-116.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited patients with Stages IIIc and IV melanoma.
Pre-assignment Details: 18 were enrolled but 10 screen-failed so only 8 proceeded with the single group assignment (Vigil treatment).
Groups:
- Vigil™ Vaccine: Autologous Vigil™ vaccine will be supplied by Gradalis, Inc. Patients will receive 1 x 10e7 cells via intradermal injection one day each month for a minimum maximum of 12 doses as long as subject is clinically stable.
  Vigil™ Vaccine
Period: Overall Study
Arm/Group | Vigil™ Vaccine
Started | 18
Completed ("Completed" means subject had successful Vigil manufacturing and had been given all the doses.) | 2
Not Completed | 16
Not completed — Disease Progression | 6
Not completed — Screen-Failures | 10

BASELINE CHARACTERISTICS:
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  Age: 0-15 Years | 0
  Age: 16-64 Years | 9
  Age: 65 and Older Years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 18
  Black/African American | 0
  Asian | 0
  Hispanic | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Enzyme-Linked ImmunoSorbent Spot (ELISPOT)
Description: To determine if subjects will have a positive (defined as >10 ELISPOTS from baseline) immune response to Vigil. Blood was collected to compare ELISPOT results from baseline until EOT (30 days after last dose).
Time Frame: Baseline, End of Treatment (30 days after last dose) up to 12 months
Population: 18 subjects were consented but only 8 subjects were administered Vigil treatment (10 screen-failed). 7 completed treatment (ELISPOT done) while 1 subject died soon after baseline (ELISPOT not done). After 12 months, 7 subjects had positive ELISPOT response. Statistical analysis was not done. This study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 18
Participants
  ELISPOT Positive After 12 months | 7
  ELISPOT Negative After 12 months | 0
  Not Done/Died immediately after Baseline | 1
  Not Done/Screen-Failed | 10

2. Secondary Outcome: Number of Alive Subjects
Description: The survival status in patients with stages IIIc and IV melanoma treated with Vigil™ vaccine was determined by following these patients up to 3 years.
Time Frame: 3 years
Population: 18 subjects were consented but only 8 were administered Vigil treatment (10 screen-failed). These 8 subjects were followed for survival up to 3 years after Vigil treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 18
Participants
  Alive Subjects After 3 years | 1
  Dead Subjects After 3 years | 7
  Screen-Failed | 10

ADVERSE EVENTS:
Arm/Group | Vigil™ Vaccine
All-Cause Mortality (participants affected / at risk) | 15/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vigil™ Vaccine (N=18)
Soft Tissue Infection (Infections and infestations) | 1 (1) — Infection of Left Great Toe
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) — Hemorrhage from tumor nodule
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Sacral Nerve Compression secondary to Metastatic Melanoma
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) — Incarcerated Abdominal Hernia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vigil™ Vaccine (N=18)
Injection Site Reaction (General disorders) | 3 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes